CLINICAL TRIAL: NCT03757923
Title: Comparison of Metformin and Pioglitazone in Regulating Menstrual Irregularities and Hyperandrogenism
Acronym: mprmih
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Jahan Ara Ainuddin, Professor, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DowUHS3
Record Dates: First submitted 2018-07-30; First posted 2018-11-29 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Menstrual Irregularities; Hyperandrogenism
Keywords: PCO; Metformin
MeSH Terms: conditions — Menstruation Disturbances; Hyperandrogenism | interventions — Metformin; Pioglitazone

STUDY DESIGN:
Intervention Model Description: randomized controlled trail
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- metformin (Experimental): TAB METFORMIN 500mg TDS
  Interventions: Drug: TAB METFORMIN
- pioglitazone (Experimental): TAB PIOGLITAZONE 30 mg OD
  Interventions: Drug: TAB PIOGLITAZONE

INTERVENTIONS:
Drug: TAB METFORMIN — INSULIN SENSITIZING AGENTS
  Arms: metformin
Drug: TAB PIOGLITAZONE — INSULIN SENSITIZING AGENT
  Arms: pioglitazone

SUMMARY:
To compare metformin with pioglitazone in improving menstrual irregularities and hyperandrogenism in women with PCOS so that an alternate and better treatment option will be available for hyperinsulinemia in pcos patients.

DETAILED DESCRIPTION:
This study will be a prospective, randomized, open label, multicentre study. It will be carried out in outpatients department of Obstetrics and gynecology, at the Dow university of Hospital and mamji hospital Karachi.

The study period will be of 6 months. Polycystic ovarian syndrome PCOS constitute most common endocrinopathy present in 4-7% women of reproductive age. Rotterdam criteria, diagnosis of PCOS require two of the three features: oligo and/or anovulation, clinical and/or biochemical signs of hyperandrogenism and polycystic ovaries by u/s and the absence of other endocrine conditions such as hypothyroidism, cushing syndrome, congenital adrenal hyperplasia, or hyperprolactinemia.

Insulin resistance and hyperinsulinemia may play a key role in pathogenesis of this syndrome by deregulating LH secretion at central level and increased stimulation of cytochrome p450 in ovary, hyperinsulinemia also decreases the circulating concentration of SHBG and contribute to greater concentration of free androgens in blood, cut off of insulin level for insulin resistance in Pakistani population is 9.25U/ml. On basis of evidence, Insulin sensitizing agents has been recently proposed as a useful treatment option in women with pcos, which by reducing insulin resistance and hyperinsulinemia, reduce the insulin driven ovarian and adrenal hyperandrogenism usually restoring normal LH and FSH secretion and ovulatory cycles.

ELIGIBILITY:
Inclusion Criteria:

1. women of age 18-40 with primary or secondary infertility.
2. Polycystic ovarian syndrome daignosed using rotterdam criteria.
3. Not taken any medication before for PCOS.

Exclusion Criteria:

1. Women having type 1 or type 2 diabetes mellitus.
2. Abnormal kidney or liver function.
3. Hypertension or heart disease.
4. Gonadotrophin induction or ovarian drilling before will not be included in this study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2018-06-18 (Actual); Primary Completion 2018-12-17 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
HIRSUTISM | 3 months
  Hirsutism will be assessed by ferryman gallaway scoring (numerical/quantitative)
POLYCYSTIC OVARIES | 3 months
  assessment on ultrasound (qualitative-present/not present)
MENSTRUAL IRREGULARITIES | 3 months
  assessment on history(qualitative-present/not present)
BMI | 3 months
  weight and height will be combined to report BMI in kg/m2

SECONDARY OUTCOMES:
SERUM FASTING INSULIN | 3 months
  unit of measure: uIU/ml
FASTING BLOOD SUGAR | 3 months
  unit of measure:mg/dl
FREE TESTOSTERONE | 3 months
  unit of measure :nmol/l
FREE ANDROGEN INDEX | 3 months
  numerical

CONTACTS AND LOCATIONS:
Overall Officials: Bader F Zuberi, FCPS, Study Director — Dow University of Health Sciences
Locations (1):
- Dow University Hospital OJHA, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No